CLINICAL TRIAL: NCT04093336
Title: Effect of Human Umbilical Cord Mesenchymal Stem Cells(MSCs) Transplantation for on Prognosis of Acute Cerebral Infarction Patients
Brief Title: Effect of Mesenchymal Stem Cells(MSCs) Transplantation for Acute Cerebral Infarction Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-DFSC-002（V3）
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Infarction, Middle Cerebral Artery; Infarction, Anterior Cerebral Artery; Cerebral Infarction; Stroke, Ischemic; Acute Stroke; Brain Infarction; Infarction, PCA; Infarction, Posterior Circulation, Brain
Keywords: Acute cerebral infarction ,Mesenchymal Stem Cells,prognosis
MeSH Terms: conditions — Infarction, Middle Cerebral Artery; Infarction, Anterior Cerebral Artery; Cerebral Infarction; Ischemic Stroke; Stroke; Brain Infarction; Infarction, Posterior Cerebral Artery

STUDY DESIGN:
Intervention Model Description: placebo controlled, randomized, double blinded
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MSCs group (Active Comparator): The people in this group will receive intravenous MSCs 2 x 10^6/kg as a single dose and standardized treatment of acute ischemic stroke.
  Interventions: Biological: human umbilical cord mesenchymal stem cells; Other: standardized treatment
- control group (Placebo Comparator): The people in this group will receive placebo and standardized treatment of acute ischemic stroke.
  Interventions: Biological: Placebo; Other: standardized treatment

INTERVENTIONS:
Biological: human umbilical cord mesenchymal stem cells — The MSCs was intravenous transplanted to acute cerebral infarction patients as a single dose.
  Arms: MSCs group
Biological: Placebo — Placebo
  Arms: control group
Other: standardized treatment — standardized treatment

SUMMARY:
This is a placebo controlled, randomized, double blinded study including Phase 1 and Phase 2. Phase I study is a safety assessment and Phase 2 study is incline to assess effectiveness of MSCs. Potential subjects must be screened and consented before enrolled.

The primary objective of this study is to determine the effects of early intravenous infusion of allogeneic human umbilical cord mesenchymal stem cells (HucMSCs or MSCs used in the following section) for patients with acute ischemic stroke. Eligible patients will receive a single dose of MSCs or placebo within 24 hours after stroke. Patients will be followed for 2 years post infusion for safety and efficacy (change in neurological symptoms and quality of life). Assessments will occur during transplantation and at 3,7, 14 days and1,3, 6, 12, 18 and 24 months after infusions of stem cells.

DETAILED DESCRIPTION:
In Phase 1 study, the eligible patients of acute cerebral infarction within 7 days after onset will be randomized to MSCs group or control group and receive intravenous MSCs 2 x 10^6/kg or placebo as a single dose, respectively. Each group will enroll 10 patients and patients will be followed for 2 years to observe the adverse events and evaluate the safety of MSCs for acute ischemic stroke patients.

The safety and preliminary effectiveness of MSCs in the treatment of acute cerebral infarction will be summarized after all patients of Phase 1 study were followed for 3 months post infusion, and the report will be submit to the academic committee and the ethics committee to evaluate before approval to begin the Phase 2 study.

In Phase 2 study, 100 patients with acute infarction within 24 hours after onset will be enrolled and randomized to MSCs group or control group. Patients will have baseline laboratory examinations and cerebral image (MRI or CTP). Enrolled patients will receive intravenous infusion of 2*10^6/kg MSCs or placebo for a single dose and follow for 24 months to assess the adverse events, neurological functional recovery and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke;
2. Age 18~80y;
3. 4≤NIHSS score≤18（including limb score≥2）and modified Rankin scale 0-1 before this cerebral ischemic stroke;
4. patients and their families understand and will cooperate within the whole process of study, and sign informed consent;
5. any of following items：①acute cerebral infarction confirmed by cerebral CT perfusion or non-contrast computed tomographic scan < 7 days after onset or ②acute cerebral infarction confirmed by cerebral MR image < 7 days after onset

Exclusion Criteria:

1. accompanied by hematological disease, severe infection, liver dysfunction (ALT>3*ULN), kidney dysfunction (Scr >2*ULN), cardiac dysfunction (NYHA grade III or IV);
2. Disturbance of consciousness, mental illness, cognitive impairment and other diseases that may affect informed consent and evaluation of study.
3. Malignancy history or found to associate cancer after this stroke
4. Pregnant or lactating women, or women have fertility requirements within 2 years;
5. Accompanied by immunodeficiency diseases or autoimmune diseases;
6. Life expectancy is less than 2 years;
7. Participated in other clinical trial within 6 months;
8. Patients received Chinese traditional medicine after onset of this stroke;
9. Patients with allergic predisposition;
10. Mental implantation or other reasons cannot tolerate magnetic resonance imaging;
11. Cannot follow up regularly or unwilling to sign informed consent;
12. Other situations not suitable for enrollment judged by the researchers;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-01-13 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
adverse events | 24 months post transplantation
  include tumorigenesis, death, pulmonary embolism, allergy, newly cerebrovascular events and other adverse events to evaluate the safety of MSCs for acute ischemic stroke patients

SECONDARY OUTCOMES:
the National Institutes of Health Stroke Scale (NIHSS) of 3 months | 3 months post transplantation
  The NIHSS neurologic examination includes 15 individual elements that measure motor and sensory function, language and speech production, vision, level of consciousness and attention, and neglect. The scores of each element are summed (range from 0 to 42) to evaluate the severity of neurological deficits. The more higher score means the more severe neurological dysfunction.
the Barthel index (BI) of 3 months | 3 months post transplantation
  The BI (range from 0 to 100) are used to assess the difference of activities of daily living between two groups. the score ≤40 means severe dependence， score 41~60 means moderate dependence, score 61~99 means mild dependence and score 100 means independence.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Li, Doctor, Principal Investigator — Shanghai East Hospital
Locations (1):
- Gang Li, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cao W, Li P. Effectiveness and Safety of Autologous Bone Marrow Stromal Cells Transplantation After Ischemic Stroke: A Meta-Analysis. Med Sci Monit. 2015 Jul 28;21:2190-5. doi: 10.12659/MSM.895081. PMID 26215395
- [Result] GBD 2013 Mortality and Causes of Death Collaborators. Global, regional, and national age-sex specific all-cause and cause-specific mortality for 240 causes of death, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Jan 10;385(9963):117-71. doi: 10.1016/S0140-6736(14)61682-2. Epub 2014 Dec 18. PMID 25530442
- [Result] Zhao Y, Yao Z, D'Souza W, Zhu C, Chun H, Zhuoga C, Zhang Q, Hu X, Zhou D. An epidemiological survey of stroke in Lhasa, Tibet, China. Stroke. 2010 Dec;41(12):2739-43. doi: 10.1161/STROKEAHA.110.586669. Epub 2010 Oct 21. PMID 20966420
- [Result] Donnan GA, Fisher M, Macleod M, Davis SM. Stroke. Lancet. 2008 May 10;371(9624):1612-23. doi: 10.1016/S0140-6736(08)60694-7. PMID 18468545
- [Result] Jauch EC, Saver JL, Adams HP Jr, Bruno A, Connors JJ, Demaerschalk BM, Khatri P, McMullan PW Jr, Qureshi AI, Rosenfield K, Scott PA, Summers DR, Wang DZ, Wintermark M, Yonas H; American Heart Association Stroke Council; Council on Cardiovascular Nursing; Council on Peripheral Vascular Disease; Council on Clinical Cardiology. Guidelines for the early management of patients with acute ischemic stroke: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Mar;44(3):870-947. doi: 10.1161/STR.0b013e318284056a. Epub 2013 Jan 31. PMID 23370205
- [Result] Campbell BC, Mitchell PJ, Kleinig TJ, Dewey HM, Churilov L, Yassi N, Yan B, Dowling RJ, Parsons MW, Oxley TJ, Wu TY, Brooks M, Simpson MA, Miteff F, Levi CR, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Priglinger M, Ang T, Scroop R, Barber PA, McGuinness B, Wijeratne T, Phan TG, Chong W, Chandra RV, Bladin CF, Badve M, Rice H, de Villiers L, Ma H, Desmond PM, Donnan GA, Davis SM; EXTEND-IA Investigators. Endovascular therapy for ischemic stroke with perfusion-imaging selection. N Engl J Med. 2015 Mar 12;372(11):1009-18. doi: 10.1056/NEJMoa1414792. Epub 2015 Feb 11. PMID 25671797
- [Result] Lee RH, Pulin AA, Seo MJ, Kota DJ, Ylostalo J, Larson BL, Semprun-Prieto L, Delafontaine P, Prockop DJ. Intravenous hMSCs improve myocardial infarction in mice because cells embolized in lung are activated to secrete the anti-inflammatory protein TSG-6. Cell Stem Cell. 2009 Jul 2;5(1):54-63. doi: 10.1016/j.stem.2009.05.003. PMID 19570514
- [Result] Crigler L, Robey RC, Asawachaicharn A, Gaupp D, Phinney DG. Human mesenchymal stem cell subpopulations express a variety of neuro-regulatory molecules and promote neuronal cell survival and neuritogenesis. Exp Neurol. 2006 Mar;198(1):54-64. doi: 10.1016/j.expneurol.2005.10.029. Epub 2005 Dec 5. PMID 16336965
- [Result] Ikeda N, Nonoguchi N, Zhao MZ, Watanabe T, Kajimoto Y, Furutama D, Kimura F, Dezawa M, Coffin RS, Otsuki Y, Kuroiwa T, Miyatake S. Bone marrow stromal cells that enhanced fibroblast growth factor-2 secretion by herpes simplex virus vector improve neurological outcome after transient focal cerebral ischemia in rats. Stroke. 2005 Dec;36(12):2725-30. doi: 10.1161/01.STR.0000190006.88896.d3. Epub 2005 Nov 10. PMID 16282547
- [Result] Ren G, Chen X, Dong F, Li W, Ren X, Zhang Y, Shi Y. Concise review: mesenchymal stem cells and translational medicine: emerging issues. Stem Cells Transl Med. 2012 Jan;1(1):51-8. doi: 10.5966/sctm.2011-0019. Epub 2011 Dec 7. PMID 23197640
- [Result] Vu Q, Xie K, Eckert M, Zhao W, Cramer SC. Meta-analysis of preclinical studies of mesenchymal stromal cells for ischemic stroke. Neurology. 2014 Apr 8;82(14):1277-86. doi: 10.1212/WNL.0000000000000278. Epub 2014 Mar 7. PMID 24610327